CLINICAL TRIAL: NCT01371968
Title: Optimal Dose of Alfentanil for Removal of Supreme Laryngeal Mask Airway During Emergence From Desflurane Anaesthesia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Malaya (Other)
Collaborators: Malaysian Society of Anaesthesiologists (Other)
Responsible Party: Principal Investigator, Lee Chew Kiok, University of Malaya, University of Malaya
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: Alfentanil LMA
Record Dates: First submitted 2011-05-04; First posted 2011-06-13 (Estimated); Last update posted 2017-10-27 (Actual); Status verified 2017-10

CONDITIONS: Airway Response
Keywords: Alfentanil; optimal dose; laryngeal mask airway
MeSH Terms: interventions — Alfentanil

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- alfentanil (Experimental): patient will received a dose of alfentanil in which the dose of alfentanil is determined by response of previously tested patient using Dixon up and down methods
  Interventions: Drug: alfentanil

INTERVENTIONS:
Drug: alfentanil — Alfentanil is administered intravenously at the end of surgery.
  Other Names: Rapifen

SUMMARY:
This study aims to determine the optimal dose of alfentanil in suppressing the airway reflexes during supreme LMA removal in anaesthetized adult.

DETAILED DESCRIPTION:
The removal of LMA may be associated with coughing, biting, agitation and airway complication such as laryngospasm. Thus it is advisable to remove the LMA when the patient is breathing spontaneously and when the airway reflexes are still depressed. A number of techniques have been used to prevent this adverse emergence phenomenon, such as removing the tube while the patient is in deep plane of anaesthesia or administration of local anaesthetic and intravenous opioids

The administration of intravenous opioids before emergence may be useful for preventing cough, agitation and hemodynamic response. Alfentanyl is proven to suppress cough and agitation during the endotracheal tube emergence. However, its use in suppressing cough in LMA patient has not been evaluated.

ELIGIBILITY:
Inclusion Criteria:

1. ASA I and II patients
2. Age 18 to 49 years old
3. Minor elective day care surgery (> 20 minute and less than 2 hours) which require local anaesthetic infiltration and does not require use of long acting opioids.

Exclusion Criteria:

1. Potential difficult airway
2. Reactive airway disease or sign and symptoms of upper respiratory tract infection.
3. History of cardiac, pulmonary and renal diseases
4. Body Mass Index > 30 kgm2.
5. Risk of aspiration.
6. Poor dentition with high risk of damage.
7. Patient refusal.

Ages: 18 Years to 49 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2011-02; Primary Completion 2011-08 (Actual); Study Completion 2011-11 (Actual)

PRIMARY OUTCOMES:
Optimal dose of alfentanil for successful LMA removal in spontaneously breathing anaesthetized adults | 6 months

SECONDARY OUTCOMES:
Number of patient with airway complication | after administration of alfentanil and within 1 min of LMA removal

CONTACTS AND LOCATIONS:
Overall Officials: Lee Chew Kiok, MBBS, Principal Investigator — Department of Anaesthesiogy, UMMC.
Locations (1):
- University Malaya Medical Centre, Kuala Lumpur, Malaysia

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol